CLINICAL TRIAL: NCT03713008
Title: Assessment of Fluid Responsiveness With Carotid Flow Change During General Anaesthesia
Brief Title: Assessment Of Carotid Flow During General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CART
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia; Fluid Responsiveness
Keywords: Fluid Responsiveness, Anesthesia, Surgery, Stroke Volume Variation, Fluid status,

STUDY DESIGN:
Intervention Model Description: All patients included in the study will receive 4 ml/kg fluid bolus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluid bolus (Experimental): Patients included in the study will receive fluid bolus.
  Interventions: Diagnostic Test: Fluid bolus

INTERVENTIONS:
Diagnostic Test: Fluid bolus — All patients included in the study will receive 5 ml/kg fluid bolus of a balanced crystalloid solution.

SUMMARY:
Proper identification of patients who would benefit from fluid infusion (fluid responsiveness) is one of the most crucial challenges in anaesthesia and critical care. Reliability of several invasive measurements used for this purpose for many years have been questioned recently. The study will evaluate consistency between carotid artery flow derivatives and standard haemodynamic measurement (LIDCO rapid) in navigation of intraoperative fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery
* Artery catheter required

Exclusion Criteria:

* Laparoscopic surgery
* Known history of carotid endarterectomy
* Known history of carotid stenosis
* Non-sinus rhythm
* Systolic or diastolic heart failure
* Chronic kidney disease
* Pulmonary hypertension
* Carotid artery anomaly
* Unable to visualise carotid artery
* Angle of correction > 60

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output | Before and 2 minutes after intervention
  A measure of change of scaled cardiac output (nCO) with LiDCO device
Change in a corrected carotid artery flow | Before and 2 minutes after intervention
  Ultrasound measure of corrected carotid artery flow time

SECONDARY OUTCOMES:
Change in pulse pressure variation | Before and 2 minutes after intervention
  A measure of change of pulse pressure variation (PPV) with LiDCO device
Change in stroke volume variation | Before and 2 minutes after intervention
  A measure of change of pulse pressure variation with LiDCO device
Change in a carotid blood flow | Before and 2 minutes after intervention
  Ultrasound measure of corrected carotid blood flow time
Change in a velocity time integral of carotid flow | Before and 2 minutes after intervention
  Ultrasound measure of velocity time integral of carotid flow
Change in the maximal systolic carotid velocity variation | Before and 2 minutes after intervention
  Ultrasound measure of the maximal systolic carotid velocity variation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Of Warsaw, Warsaw, Mazovian, Poland